CLINICAL TRIAL: NCT02173353
Title: Feasibility of Using Ultrasound to Track Respiration Motion
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, An Tai, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00020659
Record Dates: First submitted 2014-06-17; First posted 2014-06-25 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Neoplasms
Keywords: Ultrasound; Pancreatic Neoplasms; Radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pancreas cancer: Develope a stand, cradle or robotic arm to hold the ultrasound probe, to obtain an ultrasound just before a standard radiation therapy treatment is given.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound to be done just before standard radiation therapy treatment
  Other Names: Clarity

SUMMARY:
The purpose of this study is to evaluate the effectiveness of using ultrasound to image and track pancreas/duodenum motion during radiation therapy treatment delivery. Also develop a workflow and process to allow the final ultrasound system to be used routinely by radiation therapists.

DETAILED DESCRIPTION:
1. Acquire 2D and 3D ultrasound images for 5 pancreatic cancer patients using the existing Clarity system with a hand-held probe. The visibility of pancreas, duodenum, and other organs will be evaluated. Based on this image acquisition experience, design and construct stands to hold the ultrasound probe. Issues to be considered in the design include (i) avoiding the stand and probe blocking radiation beams, (ii) avoiding ultrasound going through the ribs, (iii) minimizing the effect of respiration motion. Also explore building the probe into the immobilization device (e.g., Alpha cradle) or using robotic arm.
2. Acquire ultrasound images for 20 patients with pancreatic cancer treated in the Department of Radiation Oncology department using the tools developed in Aim 1. As the standard practice, the 4 dimensional CT (4DCT) and 4 dimensional (4D) morphological and physiological MRI (T1, T2, apparent diffusion coefficient, DWI) will be acquired for treatment planning, and a respiration-gated CT will be acquired immediately before the delivery of each fraction using an in-room CT or cone-beam CT for patient positioning. The ultrasound images may be acquired during initial simulation immediately before or after the planning 4DCT and the daily gated CT, and during the treatment delivery in 2D, 3D and/or 4D modes. All raw ultrasound data will be stored.
3. Process ultrasound data acquired above to evaluate the effectiveness of using ultrasound to image and to track pancreas/duodenum motion during the treatment delivery. The images will be processed to visualize pancreas and/or surrogates, such as the boundary between pancreas and duodenum, infusion catheter. To improve the visible appearance, elastography will be explored by processing the raw data collected in Aim 2. Existing software will be used, and may be modified if necessary, to segment and to register ultrasound with CT. A tool the investigators previous develop for multimodality registration will be used to register ultrasound with MRI. Anatomic markers, such as the boundary between pancreas head and duodenum, stent, infusion catheter, may be used for registration and/or motion tracking.
4. Develop/modify workflow and process to allow the final system to be used routinely by radiation therapists. If necessary, user-friendly software tools will be developed/incorporated in the final system.
5. Explore the use of Doppler mode for tissue characterization and the potential of using it to image radiation effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will receive standard radiation therapy for pancreas cancer

Exclusion Criteria:

* Patients who will receive standard radiation therapy for sites other than pancreas cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will receive standard radiation therapy for pancreas cancer.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the use of ultrasound to detect motion of pancrease and surrounding structures | 5 years from the date of enrollment
  Design and construct stands to hold the ultrasound probe. Issues to be considered in the design include (i) avoiding the stand and probe blocking radiation beams, (ii) avoiding ultrasound going through the ribs, (iii) minimizing the effect of respiration motion. Explore building the probe into the immobilization device (e.g., Alpha cradle) or using robotic arm.

SECONDARY OUTCOMES:
Quality of ultrasound imaging for Pancreas | 3 years from the date of enrollment
  Acquire ultrasound images for 20 patients with the immobilization device (e.g., Alpha cradle) or using a robotic arm.

OTHER OUTCOMES:
Assess organ motion and compare in conjunction with magnetic resonance imaging or CT | 5 years from the date of enrollment
  Process ultrasound data acquired to evaluate the effectiveness of using ultrasound to image and to track pancreas/duodenum motion during the treatment delivery. Develop/modify workflow and process to allow the final system to be used routinely by radiation therapists. If necessary, user-friendly software tools will be developed/incorporated in the final system. Explore the use of Doppler mode for tissue characterization and the potential of using it to image radiation effects.

CONTACTS AND LOCATIONS:
Overall Officials: An Tai, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li XA, Qi XS, Pitterle M, Kalakota K, Mueller K, Erickson BA, Wang D, Schultz CJ, Firat SY, Wilson JF. Interfractional variations in patient setup and anatomic change assessed by daily computed tomography. Int J Radiat Oncol Biol Phys. 2007 Jun 1;68(2):581-91. doi: 10.1016/j.ijrobp.2006.12.024. Epub 2007 Feb 27. PMID 17331669